CLINICAL TRIAL: NCT03259100
Title: Impact of Increasing Temperature Over the Coming Century on Mortality From CVD and Stroke
Brief Title: Temperature and Mortality
Status: Completed | Type: Observational
Sponsor: Chinese Academy of Sciences (Other Government)
Responsible Party: Principal Investigator, John Speakman, Principal Investigator, Chinese Academy of Sciences
Other Study IDs: CDC and IPCC
Record Dates: First submitted 2017-08-19; First posted 2017-08-23 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: all the data collection have done by CDC. — In this study there was no intervention, just simple data collection via CDC.

SUMMARY:
The investigators evaluated the spatial association between, cardiovascular diseases (CVD) and stroke mortality rate with average ambient temperature (Ta) , and then used this relationship to model future temporal trends in mortality from CVD and stroke till the end of century (2099) using different warming scenarios across the mainland USA.

DETAILED DESCRIPTION:
the investigators used data on mortality rate (per 100,000 individuals) for CVD and stroke (between 2011 and 2013, age>35years) from the publicly available Centers for disease prevention and control (CDC) web site (www.cdc.gov). CVD mortality was defined as the number of deaths per 100,000 personyears due to circulatory causes (International Statistical Classification of Diseases, Tenth Revision, codes I00-I99).Oak Ridge National laboratory was the source of the ambient temperature data (http://www.daac.ornl.gov: files B01, B02 and C07).The investigators obtained data on prevalence of HTN (HTN was defined as systolic blood pressure (BP) of at least 140 mm Hg, self-reported use of antihypertensive treatment, or both) from county health rankings and roadmaps organisation (www.countyhealthrankings.org), which were estimated based on National Health and Nutrition Examination Survey in five two-year waves from 1999-2008 including 26,349 adults aged 30 years and older and from the Behavioral Risk Factor Surveillance System (BRFSS) from 1997-2009 including 1,283,722 adults aged 30 years and older.

ELIGIBILITY:
Inclusion Criteria:

1. age>35 years

Exclusion Criteria:

None

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We used data on mortality rate (per 100,000 individuals) for CVD and stroke (between 2011 and 2013, age>35years) from the publicly available Centers for disease prevention and control (CDC) web site (www.cdc.gov).
Sampling Method: Probability Sample
Enrollment: 17000000 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2012-01-01 (Actual); Study Completion 2013-02-01 (Actual)

PRIMARY OUTCOMES:
spatial association between, cardiovascular diseases (CVD) and stroke mortality rate with average ambient temperature | 2011-2013
  spatial association between, cardiovascular diseases (CVD) and stroke mortality rate with average ambient temperature

IPD SHARING:
Plan to Share IPD: Yes
all of our data are in public available, www.CDC.gov
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: 2011-2013
Access Criteria: there is nor criteria for the sharing these data, whole database is public access.
URL: http://www.CDC.gov

REFERENCES:
- [Background] Mazidi M, Speakman JR. Ambient particulate air pollution (PM2.5) is associated with the ratio of type 2 diabetes to obesity. Sci Rep. 2017 Aug 22;7(1):9144. doi: 10.1038/s41598-017-08287-1. PMID 28831041
- [Result] Mazidi M, Speakman JR. Higher densities of fast-food and full-service restaurants are not associated with obesity prevalence. Am J Clin Nutr. 2017 Aug;106(2):603-613. doi: 10.3945/ajcn.116.151407. Epub 2017 May 31. PMID 28566310
- [Result] Speakman JR, Heidari-Bakavoli S. Type 2 diabetes, but not obesity, prevalence is positively associated with ambient temperature. Sci Rep. 2016 Aug 1;6:30409. doi: 10.1038/srep30409. PMID 27477955
- See also: CDC website — http://www.cdc.gov